CLINICAL TRIAL: NCT03501862
Title: Mindfulness-based Interventions for People With Recent-onset Psychosis: A Randomized Controlled Trial
Brief Title: Mindfulness Intervention for People With Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Edinburgh Napier University (Other)
Responsible Party: Principal Investigator, YIP Lai King, Senior Clinical Associate, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20170811001
Record Dates: First submitted 2018-03-09; First posted 2018-04-18 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Recent-onset Psychosis
Keywords: Mindfulness; Cognitive therapy
MeSH Terms: interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: Participants referred to the study will be assessed at a screening examination to ensure eligibility and obtain written consent by a research assistant. Eligible participants will undertake a further interview on outcome measures prior to randomization within 3 weeks the commencement of intervention.
  Eligible participants will be randomly assigned to receive Mindfulness-based Cognitive Therapy for Psychosis (MBCTp) plus TAU or TAU plus Psychoeducation for Psychosis (PEp).
  Simple randomization will be used to ensure that participants will have equal opportunity to be included into the study (Altaman and Bland, 1999).
Who Masked: Outcomes Assessor
Masking Description: Assignment to the study groups will be made independently of staff involved in the recruitment and management of participants in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based intervention (Experimental): Intervention: a twelve 1.5 weekly program on mindfulness-based cognitive therapy (psychosis)
  Interventions: Behavioral: Mindfulness-based cognitive therapy (psychosis)
- Psychoeducation (Active Comparator): Intervention: a twelve 1.5 hours weekly program on psychoeducation (psychosis)
  Interventions: Behavioral: Psychoeducation (psychosis)

INTERVENTIONS:
Behavioral: Mindfulness-based cognitive therapy (psychosis) — A small group intervention is based on a structured and validated protocol that will include mindfulness practice, cognitive skills
  Arms: Mindfulness-based intervention
Behavioral: Psychoeducation (psychosis) — A small group intervention will be focusing on understanding of psychosis, treatment, relapse prevention and useful information and resources.
  Arms: Psychoeducation

SUMMARY:
People with psychosis demonstrated a tendency to use maladaptive cognitive emotion regulation strategies as compared with healthy control groups.

The present study is the first randomized controlled trial of group mindfulness-based intervention for psychosis. Half group will join the mindfulness-based cognitive intervention while another half will participate in psychoeducation to examine whether mindfulness will have a positive impact on emotion regulation and distress.

DETAILED DESCRIPTION:
Concurrently with positive and negative symptoms, affective symptoms and full affective disorder episodes are common in psychotic disorders particularly in the acute phase of illness.

Affective symptoms are a significant risk factor accounting for approximately 5-6% of suicide rates which remain or becomes higher shortly after a psychotic episode or hospital discharge (American Psychiatric Association, 2013). It has been proved that the emotion management and cognitive reappraisal were negatively associated with schizophrenia.

In the study, it is hypothesized that the intervention will have a positive impact on psychotic symptoms, general symptoms such as affective symptoms, psychological flexibility, mindfulness skills, quality of life and re-hospitalization by facilitating strategies on emotion regulation.

ELIGIBILITY:
Inclusion Criteria:

* Must be Chinese residents and aged above 18
* Have a primary diagnosis of psychosis (non-affective) and/or other psychotic disorders met the Diagnostic and Statistical Manual DSM-5
* Have been diagnosed equivalent to or less than 5 years
* Mentally stable as assessed by the researcher and a psychiatrist to comprehend the education and training provided (a pre-recruitment briefing session for potential participants will be conducted to verify their ability to follow instructions and understanding in participation, and case files will be reviewed to ensure a stable medication regime for at least 6 months) in order to ensure their ability to make a valid consent
* Able to read and understand Chinese

Exclusion Criteria:

* Have recently participated in (less than 3 months) or are receiving other structured psycho-education and/or psychotherapies
* Have comorbidities (a) developmental impairment (b) learning disability, (c) personality disorders, and/or (d) any clinically significant medical diseases (by case-file review).
* Have organic psychosis or a primary drug or alcohol addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
The Depression Anxiety Stress Scale - short form (DASS-21) | Changes will be assessed pre-study; at one week, 3-month and 6-month post-intervention
  ). It is chosen as the primary outcome measurement because scales of anxiety and depression possess the capacity to differentiate from the related state of tension and stress linking with environmental demands and emotional and physical disturbance. It is a 21-item instrument that measures over the past week symptoms of depression, anxiety and stress rated by 4-point severity or frequency scale. The scale is from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time).

SECONDARY OUTCOMES:
The Emotion Regulation Questionnaire (ERQ) | Changes will be assessed pre-study; at one week, 3-month and 6-month post-intervention
  It is a 10-item scale that was developed to measure participants' tendency to regulate their emotions in cognitive reappraisal and expressive suppression. Items are scored on a 7- point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree).
The WHOQOL-100 | Changes will be assessed pre-study; at one week, 3-month and 6-month post-intervention
  It is a self-administered questionnaire consisting of 100 items and among them, there are six domains: physical, psychological, level of independence, social relationship and environmental and spirituality.
Positive and Negative Syndrome Scale (PANSS) | Changes will be assessed pre-study; at one week, 3-month and 6-month post-intervention
  It is a 30-item, 7-point scale measuring positive and negative syndrome, differentiation of clinical symptoms and severity of illness. The seven rating points represent increasing levels of psychopathology from 1 (absent) to 7 (extreme).
Acceptance and Action Scale (AAQII) | Changes will be assessed pre-study; at one week, 3-month and 6-month post-intervention
  A seven-item questionnaire that is a commonly used self-report measure of experiential avoidance which also measures psychological inflexibility. The items are rated on a 7-point Likert scale from 1 (never true) to 7 (always true).
Five Facet Mindfulness Questionnaire (FFMQ) | Changes will be assessed pre-study; at one week, 3-month and 6-month post-intervention
  It is a 39-item self-report questionnaire that measures five facets of mindfulness: observing; describing; acting with awareness; non-judging and non-reacting. Items are scored on a 5-point Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true).
The number of re-hospitalization | It will be measured 6-month post-intervention
  To collect information from both the case files and self-reporting
The length of re-hospitalization | It will be measured 6-month post-intervention
  To collect information from both the case files and self-reporting

CONTACTS AND LOCATIONS:
Overall Officials: Thanos Karatzias, Study Director — Edinburgh Napier University
Locations (2):
- The Fourth People's Hospital, Chengdu, China
- The Society of Rehabilitation and Crime Prevention, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: SAP, CSR
Time Frame: 3-months after publication
Access Criteria: Request by sending email

DOCUMENTS (1):
  • Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT03501862/SAP_000.pdf